CLINICAL TRIAL: NCT00799227
Title: Safety and Efficacy of a New Treatment in Vitrectomized Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206207-018
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Macular Edema; Vitrectomy
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 700 µg Dexamethasone Implant (Experimental): 700 µg dexamethasone implant in the study eye at Day 1
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 700 µg Dexamethasone Posterior Segment Drug Delivery System Applicator System at Day 1 in the study eye.
  Other Names: Posurdex®; OZURDEX®

SUMMARY:
The study will evaluate the safety and efficacy of the intravitreal dexamethasone implant in the study eye of vitrectomized subjects with diabetic macular edema. Subjects will be followed for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with diabetic macular edema
* History of vitrectomy
* Central retinal thickness ≥ 275 µm
* Visual acuity between 20/320 and 20/40 in the study eye and no worse than 20/200 in the other eye

Exclusion Criteria:

* Known anticipated need for ocular surgery during the study period
* History of glaucoma or current high eye pressure requiring more than 1 medication
* Uncontrolled systemic disease
* Known allergy to the study medication
* Known steroid-responder
* Use of systemic steroids
* Female subjects that are pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Charlotte, North Carolina, United States
- Sydney, New South Wales, Australia

REFERENCES:
- [Background] Boyer DS, Faber D, Gupta S, Patel SS, Tabandeh H, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex CHAMPLAIN Study Group. Dexamethasone intravitreal implant for treatment of diabetic macular edema in vitrectomized patients. Retina. 2011 May;31(5):915-23. doi: 10.1097/IAE.0b013e318206d18c. PMID 21487341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 700 µg Dexamethasone Implant
Started | 56
Completed | 53
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | 700 µg Dexamethasone Implant
Number analyzed (Participants) | 56
Age, Customized [Number; unit: Participants]
  18 to 65 years | 37
  >65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Retinal Thickness in the Study Eye
Description: Central retinal thickness is assessed in the study eye by Optical Coherence Tomography (OCT). OCT is a laser-based, noninvasive, diagnostic system that provides high-resolution, three-dimensional images of the retina from which retinal thickness can be measured. A negative change from baseline in retinal thickness indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline, Week 26
Population: Intent to Treat: all enrolled patients
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 700 µg Dexamethasone Implant
Number analyzed (Participants) | 56
Microns
  Baseline | 403.4 (117.10)
  Change from Baseline at Week 26 | -38.9 (96.93)

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase from baseline in the number of letters read correctly indicates improvement and a decrease from baseline in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Week 26
Population: Intent to Treat: all enrolled patients
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | 700 µg Dexamethasone Implant
Number analyzed (Participants) | 56
Letters Read Correctly
  Baseline | 54.5 (12.60)
  Change from Baseline at Week 26 | 3.0 (11.11)

3. Secondary Outcome: Percentage of Patients With at Least 10 Letters of Improvement in BCVA From Baseline in the Study Eye
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Week 26
Population: Intent to treat: all enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 µg Dexamethasone Implant
Number analyzed (Participants) | 56
Percentage of Patients | 21.4

4. Secondary Outcome: Percentage of Patients With Fluorescein Leakage as Measured by Fluorescein Angiography (FA) in the Study Eye
Description: Fluorescein leakage is measured in the study eye by FA. FA is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. The assessment of fluorescein leakage compared to baseline is categorized as Improved (leakage area decreased ≥ 10%), Unchanged (leakage area changed < 10%), and Worsened (leakage area increased ≥ 10%).
Time Frame: Baseline, Week 26
Population: Intent to Treat: all enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 µg Dexamethasone Implant
Number analyzed (Participants) | 56
Percentage of Patients
  Improved at Week 26 | 33.3
  Unchanged at Week 26 | 57.1
  Worsened at Week 26 | 9.5

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs), and included all treated patients.
Arm/Group | 700 µg Dexamethasone Implant
Serious Adverse Events (participants affected / at risk) | 14/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone Implant (N=55)
Cardiac Failure Congestive (Cardiac disorders) | 2
Anoxic Encephalopathy (Nervous system disorders) | 1
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
Diabetic Foot Infection (Infections and infestations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Soft Tissue Infection (Infections and infestations) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone Implant (N=55)
Conjunctival Haemorrhage (Eye disorders) | 29
Conjunctival Hyperaemia (Eye disorders) | 11
Eye Pain (Eye disorders) | 9
Vitreous Haemorrhage (Eye disorders) | 8
Conjunctival Oedema (Eye disorders) | 7
Maculopathy (Eye disorders) | 6
Anterior Chamber Cell (Eye disorders) | 3
Foreign Body Sensation in Eyes (Eye disorders) | 3
Iritis (Eye disorders) | 3
Myodesopsia (Eye disorders) | 3
Intraocular Pressure Increased (Investigations) | 10
Renal Failure (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.